CLINICAL TRIAL: NCT03367156
Title: A Randomized Controlled Trial of Dexamethasone for Dyspnea in Cancer Patients
Brief Title: Dexamethasone in Controlling Dyspnea in Patients With Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-0591; NCI-2018-01129 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0591 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Dyspnea; Malignant Neoplasm
MeSH Terms: conditions — Dyspnea; Neoplasms | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (dexamethasone) (Experimental): Patients receive dexamethasone PO BID on days 1-28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Other: Questionnaire Administration
- Group II (placebo, dexamethasone) (Active Comparator): Patients receive placebo PO BID on days 1-14 and dexamethasone PO BID on days 15-28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (placebo, dexamethasone)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well dexamethasone works in controlling dyspnea in patients with cancer. Dexamethasone may help control dyspnea (shortness of breath) and improve lung function and quality of life in cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the intensity of dyspnea (numeric rating scale [NRS]) in the dexamethasone arm with that in the placebo arm at week 1.

SECONDARY OBJECTIVES:

I. Compare the effects of dexamethasone with those of placebo in terms of personalized dyspnea response (based on a personalized dyspnea goal), unpleasantness of dyspnea, other symptoms, health-related quality of life, respiratory physiologic function, and adverse effects at week 1 and week 2, as well as the intensity of dyspnea at week 2.

II. Identify predictive markers of dyspnea response to dexamethasone.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive dexamethasone orally (PO) twice daily (BID) on days 1-28 in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive placebo PO BID on days 1-14 and dexamethasone PO BID on days 15-28 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at days 28 and 42.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer.
* Dyspnea with an average intensity >= 4 on the dyspnea NRS (range 0-10) over the past week.
* Radiologic suspicion of thoracic involvement, such as primary or metastatic lung cancer, lymphangitic carcinomatosis, airway infiltration, lymphadenopathy, pleural or chest wall invasion.
* Seen at an outpatient clinic at MD Anderson Cancer Center or Lyndon B. Johnson (LBJ) Hospital General Oncology Clinic.
* Able to communicate in English or Spanish.
* Karnofsky performance status >= 30%.

Exclusion Criteria:

* Delirium (i.e., score > 13 on the Memorial Delirium Assessment Scale; range 1-30).
* Oxygen saturation < 90% despite supplemental oxygen > 6 L/minute.
* Previous allergic reactions to dexamethasone.
* Diagnosis of diabetes mellitus uncontrolled with oral hypoglycemic agents or insulin.
* Postsurgical open wound that has not healed at the time of enrollment.
* Any infection requiring antibiotics at the time of study enrollment.
* Major surgery within the past 2 weeks.
* Megestrol use at the time of study enrollment.
* Neutropenia (absolute neutrophil count < 1.0 x 10^9/L) at the time of study enrollment (bloodwork is not required if patient did not have chemotherapy within past 2 weeks).
* Currently receiving or expected to start cytotoxic chemotherapy or immunotherapy within 1 week of study enrollment and additional dexamethasone cannot be used concurrently as per attending oncologist.
* Severe anemia (hemoglobin < 8 g/L) not corrected prior to study enrollment (bloodwork is not required if patient did not have chemotherapy within past 2 weeks).
* Chronic obstructive pulmonary disease (COPD) exacerbation at the time of study enrollment.
* Heart failure exacerbation at the time of study enrollment.
* Expected to undergo therapeutic thoracentesis in the next 2 weeks.
* High anxiety score (>= 15/21) on the Hospital Anxiety and Depression Scale (HADS).
* Chronic systemic corticosteroid use (> 14 days) at the time of study enrollment.
* Any expected corticosteroid use during study enrollment at higher doses than will be used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Lyndon B. Johnson Hospital, Houston, Texas
  - Harris Health System Settegast Health Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hui D, Puac V, Shelal Z, Dev R, Hanneman SK, Jennings K, Ma H, Urbauer DL, Shete S, Fossella F, Liao Z, Blumenschein G Jr, Chang JY, O'Reilly M, Gandhi SJ, Tsao A, Mahler DA, Bruera E. Effect of dexamethasone on dyspnoea in patients with cancer (ABCD): a parallel-group, double-blind, randomised, controlled trial. Lancet Oncol. 2022 Oct;23(10):1321-1331. doi: 10.1016/S1470-2045(22)00508-3. Epub 2022 Sep 7. PMID 36087590
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ambulatory patients with cancer age ≥18, average dyspnea intensity over the past week ≥4/10 in a 0-10 point numeric rating scale, Karnofsky performance status ≥30% and ability to communicate in English or Spanish were selected from MD Anderson Cancer Center and Lyndon B. Johnson General Hospital, Houston, Texas, United States.
Pre-assignment Details: A total of 135 participants were enrolled but 128 were randomized. 7 participants were not randomized for various reasons.
Groups:
- Dexamethasone: Participants were given 2 capsules (4mg each) by mouth twice daily (day1-day7), then 1 capsule twice daily for the next 7 days (day 8-day 14).
- Placebo: Placebo capsules were given 2 capsules (4mg each) by mouth twice daily (day1-day7), then 1 capsule twice daily for the next 7 days (day 8-day 14).
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 85 | 43
Completed 7 Days | 76 | 38
Completed 14 Days | 61 | 35
Completed | 61 | 35
Not Completed | 24 | 8
Not completed — Lack of interest | 3 | 1
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Became ineligible | 1 | 2
Not completed — Hospitalization | 1 | 0
Not completed — Concerned about Treatment | 11 | 3
Not completed — Started new treatment | 4 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 85 | 43 | 128
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [61 to 73] | 63 [57 to 71] | 65 [60 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 24 | 74
  Male | 35 | 19 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 21
  Not Hispanic or Latino | 74 | 33 | 107
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 71 | 34 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 85 | 43 | 128
Cancer Stage [Count of Participants; unit: Participants] — Stage IV has the worst outcome.
  Participants
    Stage I-II | 18 | 15 | 33
    Stage III | 17 | 4 | 21
    Stage IV | 50 | 24 | 74
Cancer Type [Count of Participants; unit: Participants]
  Breast | 5 | 2 | 7
  Gastrointestinal | 6 | 7 | 13
  Genitourinary | 2 | 4 | 6
  Respiratory | 65 | 27 | 92
  Other | 7 | 3 | 10
Comorbidity [Count of Participants; unit: Participants]
  COPD | 32 | 12 | 44
  Asthma | 6 | 5 | 11
  Bronchiectasis | 1 | 1 | 2
  Heart Failure | 5 | 3 | 8
  Pulmonary Embolism | 2 | 1 | 3
  Other | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Dyspnea Numeric Score Over the Past 24 Hours for Baseline and Day 7 Average Intensity
Description: The average dyspnea intensity over the past 24 hours was assessed daily using a validated numeric rating scale from 0 to 10. The total score ranged from 0-10 where higher scores indicate worse dyspnea. The change in Dyspnea scores between Baseline and Day 7 were measured. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 7
Population: The Dyspnea Average Intensity Numeric score was missing for 4 participants in the Dexamethasone Arm and 1 participant in the Placebo Arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Dexamethasone; Placebo: Participants were given 2capsules (4mg each) twice daily (Day1-Day7), then 1 capsule twice daily for the next 7 days (Day 8-Day14).
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 72 | 37
score on a scale | -1.6 [-2.0 to -1.2] | -1.6 [-2.3 to -0.9]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p = 0.48, Linear Model; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.8 to 0.7]

2. Secondary Outcome: Change in Dyspnea Numeric Score Over the Past 24 Hours for Baseline and Day 14 Average Intensity
Description: The average dyspnea intensity over the past 24 hours was assessed daily using a validated numeric rating scale from 0 to 10. The total score ranged from 0-10 where higher scores indicate worse dyspnea. The change in Dyspnea scores between Baseline and Day 14 were measured. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 14
Population: Participants who were on the study at day 14 and received assessment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 68 | 35
score on a scale | -1.8 [-2.2 to -1.3] | -1.9 [-2.6 to -1.2]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p > 0.99, Linear Model; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.7 to 1]

3. Secondary Outcome: Change in Dyspnea Numeric Score Over the Past 24 Hours for Baseline and Day 7 Average Unpleasantness
Description: The average dyspnea unpleasantness over the past 24 hours was assessed daily using a validated numeric rating scale from 0 to 10. The total score ranged from 0-10 where higher scores indicate worse dyspnea. The change in Dyspnea unpleasantness scores between Baseline and Day 7 were measured. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 7
Population: The Dyspnea Average Unpleasantness Numeric score was missing for 4 participants in the Dexamethasone Arm and 2 participant in the Placebo Arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 72 | 36
score on a scale | -1.8 [-2.3 to -1.2] | -2.2 [-3.2 to -1.2]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p = 0.97, Linear Model; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.7 to 1.6]

4. Secondary Outcome: Change in Edmonton Symptom Assessment Scale (ESAS) Dyspnea Score Between Baseline and Day 7
Description: ESAS (Edmonton Symptom Assessment Scale) is a validated scale ranging from 0 (not at all) to 10 (very much) used to assess 10 symptoms commonly experienced by cancer patients during the previous 24 hours: pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep and feeling of well being. The change in ESAS fatigue score between Baseline and Day 7 were measured. Total ESAS fatigue score ranged from 0-10, with a higher score indicating higher fatigue. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 7
Population: The ESAS Dyspnea Numeric score was missing for 3 participants in the Dexamethasone Arm and 2 participant in the Placebo Arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 73 | 36
score on a scale | -1 [-3 to -1] | -1.5 [-3 to 0]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p = 0.78, Linear Model; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0]

5. Secondary Outcome: Change in European Organization for Research and Treatment of Cancer-Quality of Life (EORTC QLQ-C30) Dyspnea Score Between Baseline and Day 7
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) is a well-validated quality-of-life assessment for patients with cancer, consisting of 30 questions that encompass three symptom scales (pain, fatigue, and nausea/vomiting) and six questions about single symptoms, as well as five functional scales (physical, cognitive, role, emotional, and social) and one scale assessing global health status/quality of life. Each single symptoms have four response categories (1=not at all, and 4=very much). The change in EORTC fatigue score between Baseline and Day 7 were measured. Total scores using a complex scoring procedures ranges from 0 to 100 with a higher scores indicating higher fatigue. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 7
Population: The EORTC QLQ-C30 Dyspnea score was missing for 4 participants in the Dexamethasone Arm and 2 participant in the Placebo Arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 72 | 36
score on a scale | -33.3 [-33.3 to 0] | -33.3 [-33.3 to 0]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p = 0.93, Linear Model; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-10.6 to 9.6]

6. Secondary Outcome: Change in Dyspnea Numeric Score Over the Past 24 Hours for Baseline and Day 14 Average Unpleasantness
Description: The average dyspnea unpleasantness over the past 24 hours was assessed daily using a validated numeric rating scale from 0 to 10. The total score ranged from 0-10 where higher scores indicate worse dyspnea. The change in Dyspnea unpleasantness scores between Baseline and Day 14 were measured. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 14
Population: The Dyspnea Average Unpleasantness score was missing for 1 participant in the Placebo Arm. Participants who were on the study at day 14 and received assessment in the Dexamethasone Arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 68 | 34
score on a scale | -1.7 [-2.4 to -1.1] | -2.3 [-3.4 to -1.3]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p = 0.93, Linear Model; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.6 to 1.8]

7. Secondary Outcome: Change in Edmonton Symptom Assessment Scale (ESAS) Dyspnea Score Between Baseline and Day 14
Description: ESAS (Edmonton Symptom Assessment Scale) is a validated scale ranging from 0 (not at all) to 10 (very much) used to assess 10 symptoms commonly experienced by cancer patients during the previous 24 hours: pain, fatigue, nausea, depression, anxiety, drowsiness, dyspnea, anorexia, sleep and feeling of well being. The change in ESAS fatigue score between Baseline and Day 14 were measured. Total ESAS fatigue score ranged from 0-10, with a higher score indicating higher fatigue. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 14
Population: The ESAS Dyspnea score was missing for 3 participants in the Dexamethasone Arm and 2 participant in the Placebo Arm. Participants who were on the study at day 14 and received assessment in the Dexamethasone Arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 65 | 33
score on a scale | -2 [-3 to 0] | -1 [-4 to 0]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p = 0.82, Linear Model; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.9 to 1.1]

8. Secondary Outcome: Change in European Organization for Research and Treatment of Cancer Quality of Life (EORTC) Dyspnea Score Between Baseline and Day 14
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) is a well-validated quality-of-life assessment for patients with cancer, consisting of 30 questions that encompass three symptom scales (pain, fatigue, and nausea/vomiting) and six questions about single symptoms, as well as five functional scales (physical, cognitive, role, emotional, and social) and one scale assessing global health status/quality of life. Each single symptoms have four response categories (1=not at all, and 4=very much). The change in EORTC fatigue score between Baseline and Day 14 were measured. Total scores using a complex scoring procedures ranges from 0 to 100 with a higher scores indicating higher fatigue. Linear model analysis was used for analysis.
Time Frame: Baseline and Day 14
Population: The EORTC Dyspnea score was missing for 2 participants in the Dexamethasone Arm and 3 participant in the Placebo Arm. Participants who were on the study at day 14 and received assessment in the Dexamethasone Arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 66 | 32
score on a scale | -33.3 [-33.3 to 0] | -33.3 [-33.3 to 0]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Test type: Other; p = 0.38, Linear Model; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-17.9 to 6.9]

ADVERSE EVENTS:
Time Frame: Day 0 to Day 14
Arm/Group | Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 2/85 | 0/43
Serious Adverse Events (participants affected / at risk) | 24/85 | 3/43
Other Adverse Events (participants affected / at risk) | 32/85 | 7/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone (N=85) | Placebo (N=43)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Catheter related infection (Renal and urinary disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 0
Dehydration (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Myocardial Infarction (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pyschosis (Psychiatric disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Thromboembolic Event (Cardiac disorders) | 2 | 0
Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone (N=85) | Placebo (N=43)
Insomnia (Nervous system disorders) | 7 | 1
Pain (Nervous system disorders) | 2 | 1
Neuropsychiatric symptoms (Nervous system disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Infection (General disorders) | 9 | 3
Fatigue (General disorders) | 3 | 0
Hypertension (Cardiac disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03367156/Prot_SAP_000.pdf